CLINICAL TRIAL: NCT07146230
Title: The Selective Personalized Radio-Immunotherapy for Locally Advanced NSCLC Trial 2 (SPRINT 2)
Brief Title: The Selective Personalized Radio-Immunotherapy for Locally Advanced Non-Small Cell Lung Cancer Trial 2
Acronym: SPRINT 2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-15810
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Immunotherapy; Radiotherapy; Patient reported outcomes; Biomarkers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; monalizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Durvalumab + Monalizumab Arm (Experimental): Durvalumab 1500 mg IV and monalizumab 1500 mg IV on day 1 of a 28-day cycle for two cycles, followed by four weeks of risk adapted, dose-painted, radiotherapy, followed by durvalumab 1500 mg IV and monalizumab 1500 mg IV on day 1 of 28-day cycle for up to ten cycles.
  Interventions: Drug: Durvalumab; Drug: Monalizumab; Radiation: Radiotherapy
- Durvalumab + Oleclumab Arm (Experimental): Durvalumab 1500 mg IV on day 1 and oleclumab 3000 mg IV on day 1 and 15 of a 28-day cycle for two cycles, followed by four weeks risk adapted, dose-painted radiotherapy, followed by durvalumab 1500 mg and oleclumab 3000 mg on day 1 of 28-day cycles for up to ten cycles.
  Interventions: Drug: Durvalumab; Drug: Oleclumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is a human mAb of the immunoglobulin G 1 kappa subclass that blocks the interaction of PD-L1 (but not PD-L2) with PD 1 on T cells and CD80 (B7.1) on immune cells.
Drug: Monalizumab — Monalizumab is a humanized mAb of the IgG4 subtype that specifically binds and inhibits Cluster of Differentiation 94 (CD94)/NK cell protein group 2 A(NKG2A).
  Arms: Durvalumab + Monalizumab Arm
Drug: Oleclumab — Oleclumab is a human IgG1λ mAb that selectively binds to and inhibits the ectonucleotidase activity of CD73.
  Arms: Durvalumab + Oleclumab Arm
Radiation: Radiotherapy — PET based dose painted radiotherapy. If these treatment techniques are not available for some reason treatment may be delivered using a sequential boost technique (2.75 Gy x 17 to the low-risk PTV followed by 2.75 Gy x 3 to the high-risk planning target volume).

SUMMARY:
This is a randomized trial evaluating the efficacy and safety of sequential dual-agent immunotherapy and risk-adapted radiotherapy for patients with locally advanced non-small cell lung cancer (NSCLC) with a PD-L1 tumor proportion score of at least 50%. Participants will be randomized between two dual-agent immunotherapy regimens: durvalumab + monalizumab versus durvalumab + oleclumab.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death worldwide, with more than 1.5 million deaths per year. Non-small-cell lung cancer (NSCLC) represents more than 80% of lung cancers, and approximately one-third of NSCLC patients present with stage III disease. Locally advanced non-small cell lung carcinoma (LA-NSCLC) includes stage III NSCLC and unresectable stage II NSCLC. For several decades, standard treatment for patients with LA-NSCLC consisted of conventionally fractionated (1.8-2.0 Gy/day) radiotherapy to a total dose of approximately 60 Gy with concurrent chemotherapy. Based on the pivotal PACIFIC trial (NCT02125461), patients without disease progression after concurrent chemoradiotherapy are typically offered a one-year course of adjuvant durvalumab, which is an inhibitor of PD-L1. This "one-size-fits-all" approach has several limitations:

* Concurrent chemotherapy causes acute and subacute toxicities, which include esophagitis and pneumonitis. These adverse events impact patients' quality-of-life and can disrupt the planned treatment course, leading to increased risk of disease progression and death. Of note, approximately 25% of LA-NSCLC patients who receive chemoradiotherapy never initiate adjuvant durvalumab due to chemoradiotherapy toxicities or early disease progression. This is a major limitation of the PACIFIC approach, as immunotherapy is the most effective systemic therapy for NSCLC patients with high PD-L1 expression.
* Standard thoracic radiotherapy for LA-NSCLC delivers a uniform radiotherapy dose to the primary lung tumor and involved regional lymph nodes. Based on patterns-of-failure analyses and recent prospective trials, lower radiotherapy doses can be utilized to control small lung tumors and malignant lymph nodes. Unnecessary utilization of high-dose radiotherapy for small tumors and lymph nodes places patients at increased risk for the toxicities described above and can also cause cardiac toxicity and immunosuppression.
* For many patients, deferring immunotherapy for LA-NSCLC until after completion of chemoradiotherapy is problematic. As recently demonstrated in a randomized trial comparing preoperative immunotherapy to postoperative immunotherapy for melanoma, immunotherapy is most effective when utilized to treat intact tumors in patients with preserved immune systems. The current practice of employing regional lymph node irradiation prior to immunotherapy for LA-NSCLC appears to be particularly deleterious. As mentioned above, some LA-NSCLC patients who start treatment with chemoradiotherapy never reach the key phase of adjuvant immunotherapy.

To address the limitations described above and improve the safety and efficacy of LA-NSCLC therapy, Montefiore-Einstein has led a series of trials testing more personalized treatment approaches. The Selective Personalized RadioImmunotherapy for Locally Advanced NSCLC Trial (SPRINT, NCT03523702), tested a novel chemotherapy-free approach where 25 LA-NSCLC patients with PD-L1 TPS ≥ 50% were treated with three cycles of induction pembrolizumab, followed by a four-week course of risk-adapted and de-intensified thoracic radiotherapy based on restaging PET/CT, followed by consolidation pembrolizumab to complete a one-year treatment course. Patients with PD-L1 TPS < 50% could be enrolled and treated with standard concurrent chemoradiotherapy followed by standard adjuvant therapy.

Study participants will receive two cycles of dual-agent immunotherapy followed by a four-week course of risk-adapted radiotherapy, followed by up to ten cycles of dual-agent immunotherapy. Subjects who discontinue study therapy due to disease progression or treatment intolerance may receive additional therapy, at the discretion of the treating physicians.

Durvalumab is a human monoclonal antibody (mAb) of the immunoglobulin G 1 kappa subclass that blocks the interaction of PD-L1 (but not PD-L2) with PD 1 on T cells and CD80 (B7.1) on immune cells. It has been developed by AstraZeneca for use in the treatment of cancer. The mechanism of action for durvalumab is interference in the interaction of PD-L1 with PD 1 and CD80 (B7-1). Blockade of PD-L1/PD-1 and PD-L1/CD80 interactions releases the inhibition of immune responses, including those that may result in tumor elimination. In vitro studies demonstrate that durvalumab antagonizes the inhibitory effect of PD-L1 on primary human T cells, resulting in the restored proliferation of interferon-γ (IFN-γ). In vivo studies have shown that durvalumab inhibits tumor growth in xenograft models via a T cell dependent mechanism. Based on these data, durvalumab is expected to stimulate the participant's antitumor immune response by binding to PD-L1 and shifting the balance toward an antitumor response. Durvalumab has been engineered to reduce antibody dependent cellular cytotoxicity and complement-dependent cytotoxicity.

To date, durvalumab has been given to thousands of participants as part of ongoing studies either as monotherapy or in combination with other anticancer agents.

Durvalumab is approved in some countries as monotherapy for unresectable Stage III NSCLC (following chemoradiation therapy), and in combination with chemotherapy for extensive stage small cell lung cancer and for locally advanced or metastatic biliary tract cancer. Durvalumab is approved as monotherapy in unresectable hepatocellular carcinoma in Japan. Durvalumab is also approved when administered in combination with tremelimumab for unresectable hepatocellular carcinoma, and also in combination with tremelimumab plus chemotherapy for participants with metastatic NSCLC without epidermal growth factor receptor (EGFR) or Anaplastic Lymphoma Kinase (ALK) mutations.

A fixed dosing approach is preferred by the prescribing community due to ease of use and reduced dosing errors. Given the expectation of similar pharmacokinetic (PK) exposure and variability, AstraZeneca considered it feasible to switch to fixed dosing regimens.

A fixed dose of 1500 mg durvalumab administered q4w is to be used for all participants with a body weight greater than 30 kg. Currently, the use of a fixed dose of 1500 mg durvalumab, administered both in combination with chemotherapy and as monotherapy, is approved for treatment of extensive stage small cell lung cancer. Additionally, the 1500 mg fixed dose is approved in some regions as monotherapy for unresectable stage III NSCLC.

For participants in this study, who will have locally advanced NSCLC with high PD-L1 expression, durvalumab is expected to be among the most effective systemic treatment options to reduce the risk of disease progression and death. The researchers believe that initiation of durvalumab prior to receipt of thoracic radiotherapy, which will take place in this study, will yield greater benefits than what is observed when durvalumab is planned as adjuvant therapy after chemoradiotherapy. One reason is that durvalumab may be more effective when given to patients with intact immune systems. Chemoradiotherapy is known to cause lymphopenia, which has been associated with reduced efficacy of immunotherapy and inferior clinical outcomes. Additionally, administration of durvalumab prior to radiotherapy can reduce participants' thoracic disease burden, which will reduce the required extent of thoracic irradiation and should reduce the risk of acute and long-term treatment toxicity.

Monalizumab is a humanized mAb of the IgG4 subtype that specifically binds and inhibits Cluster of Differentiation 94 (CD94)/NK cell protein group 2 A(NKG2A). Engagement of NKG2A, a receptor found on both the natural killer and CD8+ T cells, culminates in inhibition of immune cell effector functions. As a heterodimer with CD94 on the cell surface, NKG2A can recognize the non-classical major histocompatibility complex molecules, human leukocyte antigen (HLA)-E expressed by antigen presenting cells. HLA-E has been shown to be overexpressed in various tumor types, including lung cancer. This overexpression functions as a negative prognostic factor in the lung carcinoma. These findings suggest that unleashing NK cell and CD8+ T cell activity by inhibiting NKG2A/HLA-E binding in lung cancer may contribute to stronger anti-tumor immunity.

Oleclumab is a human IgG1λ mAb that selectively binds to and inhibits the ectonucleotidase activity of CD73. Oleclumab inhibits the production of adenosine and inorganic phosphate from adenosine monophosphate (AMP) by CD73. Adenosine creates an immunosuppressive tumor microenvironment by impairing the proliferation of effector cytotoxic cells and promoting generation of immunosuppressive regulatory T cells, myeloid derived suppressor cells and tumor associated macrophages. In NSCLC, high expression of CD73 has been associated with poor prognosis.

The addition of monalizumab to adjuvant durvalumab after chemoradiotherapy, as well as the addition of oleclumab to adjuvant durvalumab after chemotherapy, for patients with LA-NSCLC improved PFS rates in the COAST trial (NCT03822351). PACIFIC-9 trial (NCT05221840) is an ongoing confirmatory phase III study testing the same approaches. The combination of durvalumab and monalizumab, as well as the combination of durvalumab an oleclumab, were tested as neoadjuvant therapies before surgery in the NeoCOAST trial (NCT03794544), where these combination therapies each numerically improved pathologic response rates compared to durvalumab alone. Of note, results from both COAST and NeoCOAST suggest that the additions of monalizumab to durvalumab, and of oleclumab to durvalumab, did not increase toxicity rates. There, existing data support testing monalizumab in combination with durvalumab, and oleclumab in combination with durvalumab, as induction therapies before definitive radiotherapy and as consolidation therapies after radiotherapy, to reduce the extent of thoracic irradiation required and improve local and distant disease control.

For this study, participants will undergo standard evaluations, including biopsy and PD-L1 testing, staging positron emission tomography/computed tomography (PET/CT), and laboratory studies, before treatment. PET/CT will be performed after induction immunotherapy for biologic response assessment and to aid with radiotherapy planning. CT will be performed after radiotherapy and then approximately every three months throughout the first year of study participation. Subsequent tumor assessments will follow institutional standards. Safety will be assessed throughout using Common Terminology Criteria for Adverse Events (CTCAE).

The researchers believe that, for patients with locally advanced NSCLC with PD-L1 tumor proportion score of at least 50%, sequential treatment with dual-agent immunotherapy and risk-adapted radiotherapy will be safe and effective. The specific hypothesis that will be tested as the primary objective of this study is that induction dual-agent immunotherapy will yield response rates that are higher than what had been observed in a previous trial with single-agent immunotherapy. These response rates will be assessed using Fludeoxyglucose (18F)-positron emission tomography (FDG-PET) imaging, as response on PET to induction therapy was identified as a powerful predictor of long-term clinical outcomes in the previous trial.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Patient is willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations, including follow-up.
3. Age > 18 years at time of study entry
4. Body weight ≥35 kg
5. Life expectancy of at least 12 weeks
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Previously untreated, pathologically proven NSCLC and one of the following stages:

   1. American Joint Committee on Cancer (AJCC) version 8 Stage II disease, medically or technically unresectable
   2. AJCC version 8 Stage III disease
   3. Recurrent disease after curative-intent treatment for early-stage NSCLC, with current disease burden that would qualify as AJCC version 8 stage II-III
8. PD-L1 testing performed using an FDA-approved immunohistochemical assay and demonstrating tumor proportion score (TPS) of at least 50%.
9. Whole body PET/CT within 42 days prior to study entry demonstrating at least one hypermetabolic pulmonary lesion or thoracic lymph node.
10. MRI of the brain or head CT with contrast within 42 days prior to study entry.
11. PFTs within 42 days of study entry are recommended but not required.
12. Adequate normal organ and marrow function as defined below:

Hemoglobin ≥9.0 g/dL Absolute neutrophil count (ANC) ≥ 1.5 × 109 /L Platelet count ≥75 × 109/L Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with Gilbert's syndrome.

Serum albumin ≥ 3.0 g/dL AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal Measured creatinine clearance >40 mL/min or Calculated creatinine clearance >40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.

* Males: (Weight in kg) x (140 - Age) ÷ (72 x serum creatinine in mg/dL)
* Females: (Weight in kg) x (140 - Age) x 0.85 ÷ (72 x serum creatinine in mg/dL)

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 months
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
3. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy, with these exceptions:

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment on this study may be included after consultation with the Study Physician.
4. Any concurrent chemotherapy, Intraperitoneal (IP) chemotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. History of another primary malignancy except for

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease
6. History of leptomeningeal carcinomatosis
7. Prior radiotherapy that would preclude safe delivery of radiotherapy as specified in this study.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first planned dose of IP.
9. History of allogenic organ transplantation.
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of grade 3 or greater edema (e.g., peripheral, pulmonary)
13. History of venous thrombosis within the past 3 months prior to the planned first dose of study treatment. Note: Subjects with thrombosis due to mechanical obstruction by the tumor that is found incidentally and is asymptomatic and does not require therapy may be enrolled at the investigator's discretion and should be closely monitored.
14. Cardiac or peripheral vascular disease meeting any of the following criteria:

    1. History of myocardial infarction in the prior 12 months
    2. History of stroke or transient ischemic attack requiring medical therapy
15. Congestive heart failure ≥ Class 3 based on New York Heart Association Functional Classification
16. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
17. History of active primary immunodeficiency
18. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening.

    1. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible.
    2. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
19. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
20. Current or prior use of immunosuppressive medication within 14 days before the first dose of IP. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
21. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP.
22. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
23. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
24. Patients who have received prior anti-PD-1 or anti PD-L1 therapy:

    1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy
    2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    3. Must not have experienced a ≥Grade 3 immune related AE or an immune-related neurologic or ocular AE of any grade while receiving prior immunotherapy. Note: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Response rate observed using FDG-PET imaging | Following completion of two cycles of induction dual-agent immunotherapy; approximately 9 weeks
  Response rate will be assessed using Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) criteria prior to radiotherapy initiation. Response rate will be defined as a ≥ 30% decline in maximum standardized uptake value (SUV) without development of new disease sites. Response rates, which include partial metabolic responses and complete metabolic responses, will be presented as a count and percentage for each study arm. Participants who do not undergo FDG-PET after completion of induction immunotherapy (e.g., due to clinical disease progression, toxicity, or death) will be counted as non-responders.

SECONDARY OUTCOMES:
Response rates observed using Computed Tomography (CT) | Following completion of two cycles of induction dual-agent immunotherapy; approximately 9 weeks
  Response rates will also be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) criteria prior to radiotherapy initiation. Response rates, which include partial responses and complete responses, will be presented as a count and percentage for each study arm, along with a 95% Clopper-Pearson exact confidence interval. Participants who do not undergo imaging after completion of induction immunotherapy (e.g., due to clinical disease progression, toxicity, or death) will be counted as non-responders.
Progression free survival (PFS) | From randomization until the date of death, up to approximately 54 weeks
  PFS duration will be defined for each participant as the interval from the date of randomization to the first date of documented disease progression or death due to any cause, whichever occurs first. Subjects who die without reported progression will be considered to have the PFS event on the date of their death. Subjects who do not progress or die will be censored on the date of their last evaluable tumor assessment or clinic visit. PFS duration will be summarized for each study arm and estimated using the Kaplan-Meier product-limit method.
Overall survival (OS) rates | From randomization until the date of death, up to approximately 54 weeks
  OS duration will be defined for each participant as the interval from the date of randomization to the date of death due to any cause. Subjects who do not die will be censored on the date of their last evaluable tumor assessment or clinic visit. OS duration will be summarized for each study arm and estimated using the Kaplan-Meier method.
Rates of disease progression during treatment | Following completion of two cycles of induction dual-agent immunotherapy; approximately 9 weeks
  Rates of disease progression during induction dual-agent immunotherapy and before initiation of thoracic radiotherapy will be assessed using a binary ("Yes" or "No") outcome. PET/CT and/or biopsy to confirm disease progression may be performed, at the discretion of the treating physicians. In some cases, disease progression may be detected by other means (e.g., thoracentesis demonstrating malignant effusion). Rates of disease progression will be summarized and reported for each arm as counts and percentages.
Physician-scored adverse events | During study therapy; up to approximately 54 weeks
  Physician-scored adverse events will be scored using Common Terminology of Common Adverse Events (CTCAE) version 5.0. All Grade 2 and ≥ Grade 3 adverse events related to treatment will be summarized by study arm and presented using counts and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin R Ohri, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Bradley JD, Hu C, Komaki RR, Masters GA, Blumenschein GR, Schild SE, Bogart JA, Forster KM, Magliocco AM, Kavadi VS, Narayan S, Iyengar P, Robinson CG, Wynn RB, Koprowski CD, Olson MR, Meng J, Paulus R, Curran WJ Jr, Choy H. Long-Term Results of NRG Oncology RTOG 0617: Standard- Versus High-Dose Chemoradiotherapy With or Without Cetuximab for Unresectable Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2020 Mar 1;38(7):706-714. doi: 10.1200/JCO.19.01162. Epub 2019 Dec 16. PMID 31841363
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Machtay M, Bae K, Movsas B, Paulus R, Gore EM, Komaki R, Albain K, Sause WT, Curran WJ. Higher biologically effective dose of radiotherapy is associated with improved outcomes for locally advanced non-small cell lung carcinoma treated with chemoradiation: an analysis of the Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):425-34. doi: 10.1016/j.ijrobp.2010.09.004. Epub 2010 Oct 25. PMID 20980108
- [Background] Fowler JF, Chappell R. Non-small cell lung tumors repopulate rapidly during radiation therapy. Int J Radiat Oncol Biol Phys. 2000 Jan 15;46(2):516-7. doi: 10.1016/s0360-3016(99)00364-8. No abstract available. PMID 10661362
- [Background] Shaverdian N, Offin MD, Rimner A, Shepherd AF, Wu AJ, Rudin CM, Hellmann MD, Chaft JE, Gomez DR. Utilization and factors precluding the initiation of consolidative durvalumab in unresectable stage III non-small cell lung cancer. Radiother Oncol. 2020 Mar;144:101-104. doi: 10.1016/j.radonc.2019.11.015. Epub 2019 Nov 28. PMID 31786421
- [Background] Bruni A, Scotti V, Borghetti P, Vagge S, Cozzi S, D'Angelo E, Giaj Levra N, Fozza A, Taraborrelli M, Piperno G, Vanoni V, Sepulcri M, Trovo M, Nardone V, Lattanzi E, Bou Selman S, Bertolini F, Franceschini D, Agustoni F, Jereczek-Fossa BA, Magrini SM, Livi L, Lohr F, Filippi AR. A Real-World, Multicenter, Observational Retrospective Study of Durvalumab After Concomitant or Sequential Chemoradiation for Unresectable Stage III Non-Small Cell Lung Cancer. Front Oncol. 2021 Sep 28;11:744956. doi: 10.3389/fonc.2021.744956. eCollection 2021. PMID 34650927
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Vandormael K, Riccio A, Yang J, Pietanza MC, Brahmer JR. Updated Analysis of KEYNOTE-024: Pembrolizumab Versus Platinum-Based Chemotherapy for Advanced Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score of 50% or Greater. J Clin Oncol. 2019 Mar 1;37(7):537-546. doi: 10.1200/JCO.18.00149. Epub 2019 Jan 8. PMID 30620668
- [Background] Ohri N, Bodner WR, Halmos B, Cheng H, Perez-Soler R, Keller SM, Kalnicki S, Garg M. 18F-Fluorodeoxyglucose/Positron Emission Tomography Predicts Patterns of Failure After Definitive Chemoradiation Therapy for Locally Advanced Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2017 Feb 1;97(2):372-380. doi: 10.1016/j.ijrobp.2016.10.031. Epub 2016 Oct 26. PMID 28068244
- [Background] Ohri N, Piperdi B, Garg MK, Bodner WR, Gucalp R, Perez-Soler R, Keller SM, Guha C. Pre-treatment FDG-PET predicts the site of in-field progression following concurrent chemoradiotherapy for stage III non-small cell lung cancer. Lung Cancer. 2015 Jan;87(1):23-7. doi: 10.1016/j.lungcan.2014.10.016. Epub 2014 Nov 6. PMID 25468149
- [Background] Binkley MS, Koenig JL, Kashyap M, Xiang M, Liu Y, Sodji Q, Maxim PG, Diehn M, Loo BW Jr, Gensheimer MF. Predicting per-lesion local recurrence in locally advanced non-small cell lung cancer following definitive radiation therapy using pre- and mid-treatment metabolic tumor volume. Radiat Oncol. 2020 May 19;15(1):114. doi: 10.1186/s13014-020-01546-y. PMID 32429982
- [Background] Ohri N, Bodner WR, Kabarriti R, Shankar V, Cheng H, Abraham T, Halmos B, Gucalp R, Perez-Soler R, Kalnicki S, Garg M. Positron Emission Tomography-Adjusted Intensity Modulated Radiation Therapy for Locally Advanced Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2018 Nov 15;102(4):709-715. doi: 10.1016/j.ijrobp.2017.10.032. Epub 2017 Oct 28. PMID 29249527
- [Background] Dess RT, Sun Y, Matuszak MM, Sun G, Soni PD, Bazzi L, Murthy VL, Hearn JWD, Kong FM, Kalemkerian GP, Hayman JA, Ten Haken RK, Lawrence TS, Schipper MJ, Jolly S. Cardiac Events After Radiation Therapy: Combined Analysis of Prospective Multicenter Trials for Locally Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2017 May 1;35(13):1395-1402. doi: 10.1200/JCO.2016.71.6142. Epub 2017 Mar 16. PMID 28301264
- [Background] Wang K, Eblan MJ, Deal AM, Lipner M, Zagar TM, Wang Y, Mavroidis P, Lee CB, Jensen BC, Rosenman JG, Socinski MA, Stinchcombe TE, Marks LB. Cardiac Toxicity After Radiotherapy for Stage III Non-Small-Cell Lung Cancer: Pooled Analysis of Dose-Escalation Trials Delivering 70 to 90 Gy. J Clin Oncol. 2017 May 1;35(13):1387-1394. doi: 10.1200/JCO.2016.70.0229. Epub 2017 Jan 23. PMID 28113017
- [Background] Contreras JA, Lin AJ, Weiner A, Speirs C, Samson P, Mullen D, Campian J, Bradley J, Roach M, Robinson C. Cardiac dose is associated with immunosuppression and poor survival in locally advanced non-small cell lung cancer. Radiother Oncol. 2018 Sep;128(3):498-504. doi: 10.1016/j.radonc.2018.05.017. Epub 2018 May 30. PMID 29859754
- [Background] Chen D, Patel RR, Verma V, Ramapriyan R, Barsoumian HB, Cortez MA, Welsh JW. Interaction between lymphopenia, radiotherapy technique, dosimetry, and survival outcomes in lung cancer patients receiving combined immunotherapy and radiotherapy. Radiother Oncol. 2020 Sep;150:114-120. doi: 10.1016/j.radonc.2020.05.051. Epub 2020 Jun 7. PMID 32525003
- [Background] Tang C, Liao Z, Gomez D, Levy L, Zhuang Y, Gebremichael RA, Hong DS, Komaki R, Welsh JW. Lymphopenia association with gross tumor volume and lung V5 and its effects on non-small cell lung cancer patient outcomes. Int J Radiat Oncol Biol Phys. 2014 Aug 1;89(5):1084-1091. doi: 10.1016/j.ijrobp.2014.04.025. Epub 2014 Jul 8. PMID 25035212
- [Background] Darragh LB, Gadwa J, Pham TT, Van Court B, Neupert B, Olimpo NA, Nguyen K, Nguyen D, Knitz MW, Hoen M, Corbo S, Joshi M, Zhuang Y, Amann M, Wang XJ, Dow S, Kedl RM, Samedi V, Boss MK, Karam SD. Elective nodal irradiation mitigates local and systemic immunity generated by combination radiation and immunotherapy in head and neck tumors. Nat Commun. 2022 Nov 16;13(1):7015. doi: 10.1038/s41467-022-34676-w. PMID 36385142
- [Background] Ohri N, Jolly S, Cooper BT, Kabarriti R, Bodner WR, Klein J, Guha C, Viswanathan S, Shum E, Sabari JK, Cheng H, Gucalp RA, Castellucci E, Qin A, Gadgeel SM, Halmos B. Selective Personalized RadioImmunotherapy for Locally Advanced Non-Small-Cell Lung Cancer Trial (SPRINT). J Clin Oncol. 2024 Feb 10;42(5):562-570. doi: 10.1200/JCO.23.00627. Epub 2023 Nov 21. PMID 37988638
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Background] Basch E, Becker C, Rogak LJ, Schrag D, Reeve BB, Spears P, Smith ML, Gounder MM, Mahoney MR, Schwartz GK, Bennett AV, Mendoza TR, Cleeland CS, Sloan JA, Bruner DW, Schwab G, Atkinson TM, Thanarajasingam G, Bertagnolli MM, Dueck AC. Composite grading algorithm for the National Cancer Institute's Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). Clin Trials. 2021 Feb;18(1):104-114. doi: 10.1177/1740774520975120. Epub 2020 Dec 1. PMID 33258687
- [Background] Basch E, Reeve BB, Mitchell SA, Clauser SB, Minasian LM, Dueck AC, Mendoza TR, Hay J, Atkinson TM, Abernethy AP, Bruner DW, Cleeland CS, Sloan JA, Chilukuri R, Baumgartner P, Denicoff A, St Germain D, O'Mara AM, Chen A, Kelaghan J, Bennett AV, Sit L, Rogak L, Barz A, Paul DB, Schrag D. Development of the National Cancer Institute's patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE). J Natl Cancer Inst. 2014 Sep 29;106(9):dju244. doi: 10.1093/jnci/dju244. Print 2014 Sep. PMID 25265940
- [Background] Stewart R, Morrow M, Hammond SA, Mulgrew K, Marcus D, Poon E, Watkins A, Mullins S, Chodorge M, Andrews J, Bannister D, Dick E, Crawford N, Parmentier J, Alimzhanov M, Babcook JS, Foltz IN, Buchanan A, Bedian V, Wilkinson RW, McCourt M. Identification and Characterization of MEDI4736, an Antagonistic Anti-PD-L1 Monoclonal Antibody. Cancer Immunol Res. 2015 Sep;3(9):1052-62. doi: 10.1158/2326-6066.CIR-14-0191. Epub 2015 May 5. PMID 25943534
- [Background] Narwal R, Roskos LK, Robbie GJ. Population pharmacokinetics of sifalimumab, an investigational anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus. Clin Pharmacokinet. 2013 Nov;52(11):1017-27. doi: 10.1007/s40262-013-0085-2. PMID 23754736
- [Background] Ng CM, Lum BL, Gimenez V, Kelsey S, Allison D. Rationale for fixed dosing of pertuzumab in cancer patients based on population pharmacokinetic analysis. Pharm Res. 2006 Jun;23(6):1275-84. doi: 10.1007/s11095-006-0205-x. Epub 2006 May 26. PMID 16715358
- [Background] Wang DD, Zhang S, Zhao H, Men AY, Parivar K. Fixed dosing versus body size-based dosing of monoclonal antibodies in adult clinical trials. J Clin Pharmacol. 2009 Sep;49(9):1012-24. doi: 10.1177/0091270009337512. Epub 2009 Jul 20. PMID 19620385
- [Background] Zhang S, Shi R, Li C, Parivar K, Wang DD. Fixed dosing versus body size-based dosing of therapeutic peptides and proteins in adults. J Clin Pharmacol. 2012 Jan;52(1):18-28. doi: 10.1177/0091270010388648. Epub 2011 Jan 13. PMID 21233304
- [Background] Shiraishi Y, Fang P, Xu C, Song J, Krishnan S, Koay EJ, Mehran RJ, Hofstetter WL, Blum-Murphy M, Ajani JA, Komaki R, Minsky B, Mohan R, Hsu CC, Hobbs BP, Lin SH. Severe lymphopenia during neoadjuvant chemoradiation for esophageal cancer: A propensity matched analysis of the relative risk of proton versus photon-based radiation therapy. Radiother Oncol. 2018 Jul;128(1):154-160. doi: 10.1016/j.radonc.2017.11.028. Epub 2017 Dec 14. PMID 29248170
- [Background] Abravan A, Faivre-Finn C, Kennedy J, McWilliam A, van Herk M. Radiotherapy-Related Lymphopenia Affects Overall Survival in Patients With Lung Cancer. J Thorac Oncol. 2020 Oct;15(10):1624-1635. doi: 10.1016/j.jtho.2020.06.008. Epub 2020 Jun 14. PMID 32553694
- [Background] Friedes C, Chakrabarti T, Olson S, Prichett L, Brahmer JR, Forde PM, Voong RK, Marrone KA, Lam VK, Hann CL, Broderick SR, Battafarano RJ, Ha JS, Bush EL, Yang SC, Hales RK, Feliciano JL. Association of severe lymphopenia and disease progression in unresectable locally advanced non-small cell lung cancer treated with definitive chemoradiation and immunotherapy. Lung Cancer. 2021 Apr;154:36-43. doi: 10.1016/j.lungcan.2021.01.022. Epub 2021 Jan 27. PMID 33611224
- [Background] Le Drean E, Vely F, Olcese L, Cambiaggi A, Guia S, Krystal G, Gervois N, Moretta A, Jotereau F, Vivier E. Inhibition of antigen-induced T cell response and antibody-induced NK cell cytotoxicity by NKG2A: association of NKG2A with SHP-1 and SHP-2 protein-tyrosine phosphatases. Eur J Immunol. 1998 Jan;28(1):264-76. doi: 10.1002/(SICI)1521-4141(199801)28:013.0.CO;2-O. PMID 9485206
- [Background] McMahon CW, Raulet DH. Expression and function of NK cell receptors in CD8+ T cells. Curr Opin Immunol. 2001 Aug;13(4):465-70. doi: 10.1016/s0952-7915(00)00242-9. PMID 11498303
- [Background] Navarro F, Llano M, Bellon T, Colonna M, Geraghty DE, Lopez-Botet M. The ILT2(LIR1) and CD94/NKG2A NK cell receptors respectively recognize HLA-G1 and HLA-E molecules co-expressed on target cells. Eur J Immunol. 1999 Jan;29(1):277-83. doi: 10.1002/(SICI)1521-4141(199901)29:013.0.CO;2-4. PMID 9933109
- [Background] Talebian Yazdi M, van Riet S, van Schadewijk A, Fiocco M, van Hall T, Taube C, Hiemstra PS, van der Burg SH. The positive prognostic effect of stromal CD8+ tumor-infiltrating T cells is restrained by the expression of HLA-E in non-small cell lung carcinoma. Oncotarget. 2016 Jan 19;7(3):3477-88. doi: 10.18632/oncotarget.6506. PMID 26658106
- [Background] Platonova S, Cherfils-Vicini J, Damotte D, Crozet L, Vieillard V, Validire P, Andre P, Dieu-Nosjean MC, Alifano M, Regnard JF, Fridman WH, Sautes-Fridman C, Cremer I. Profound coordinated alterations of intratumoral NK cell phenotype and function in lung carcinoma. Cancer Res. 2011 Aug 15;71(16):5412-22. doi: 10.1158/0008-5472.CAN-10-4179. Epub 2011 Jun 27. PMID 21708957
- [Background] Herbst RS, Majem M, Barlesi F, Carcereny E, Chu Q, Monnet I, Sanchez-Hernandez A, Dakhil S, Camidge DR, Winzer L, Soo-Hoo Y, Cooper ZA, Kumar R, Bothos J, Aggarwal C, Martinez-Marti A. COAST: An Open-Label, Phase II, Multidrug Platform Study of Durvalumab Alone or in Combination With Oleclumab or Monalizumab in Patients With Unresectable, Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Oct 10;40(29):3383-3393. doi: 10.1200/JCO.22.00227. Epub 2022 Apr 22. PMID 35452273
- [Background] Antonioli L, Blandizzi C, Pacher P, Hasko G. Immunity, inflammation and cancer: a leading role for adenosine. Nat Rev Cancer. 2013 Dec;13(12):842-57. doi: 10.1038/nrc3613. Epub 2013 Nov 14. PMID 24226193
- [Background] Gotay CC, Kawamoto CT, Bottomley A, Efficace F. The prognostic significance of patient-reported outcomes in cancer clinical trials. J Clin Oncol. 2008 Mar 10;26(8):1355-63. doi: 10.1200/JCO.2007.13.3439. Epub 2008 Jan 28. PMID 18227528
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Fogh SE, Deshmukh S, Berk LB, Dueck AC, Roof K, Yacoub S, Gergel T, Stephans K, Rimner A, DeNittis A, Pablo J, Rineer J, Williams TM, Bruner D. A Randomized Phase 2 Trial of Prophylactic Manuka Honey for the Reduction of Chemoradiation Therapy-Induced Esophagitis During the Treatment of Lung Cancer: Results of NRG Oncology RTOG 1012. Int J Radiat Oncol Biol Phys. 2017 Mar 15;97(4):786-796. doi: 10.1016/j.ijrobp.2016.11.022. Epub 2016 Nov 23. PMID 28244415
- [Background] Ohri N, Kabarriti R, Bodner WR, Mehta KJ, Shankar V, Halmos B, Haigentz M Jr, Rapkin B, Guha C, Kalnicki S, Garg M. Continuous Activity Monitoring During Concurrent Chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2017 Apr 1;97(5):1061-1065. doi: 10.1016/j.ijrobp.2016.12.030. Epub 2016 Dec 25. PMID 28332990
- [Background] Ohri N, Halmos B, Bodner WR, Cheng H, Guha C, Kalnicki S, Garg M. Daily Step Counts: A New Prognostic Factor in Locally Advanced Non-Small Cell Lung Cancer? Int J Radiat Oncol Biol Phys. 2019 Nov 15;105(4):745-751. doi: 10.1016/j.ijrobp.2019.07.055. Epub 2019 Aug 7. PMID 31398385
- [Background] Ewald B, Duke J, Thakkinstian A, Attia J, Smith W. Physical activity of older Australians measured by pedometry. Australas J Ageing. 2009 Sep;28(3):127-33. doi: 10.1111/j.1741-6612.2009.00372.x. PMID 19845652
- [Background] Paul S, Bodner WR, Garg M, Tang J, Ohri N. Cardiac Irradiation Predicts Activity Decline in Patients Receiving Concurrent Chemoradiation for Locally Advanced Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Nov 1;108(3):597-601. doi: 10.1016/j.ijrobp.2020.05.042. Epub 2020 Jun 1. PMID 32497682
- [Background] Zelen M. The randomization and stratification of patients to clinical trials. J Chronic Dis. 1974 Sep;27(7-8):365-75. doi: 10.1016/0021-9681(74)90015-0. No abstract available. PMID 4612056
- [Background] Werner-Wasik M, Nelson AD, Choi W, Arai Y, Faulhaber PF, Kang P, Almeida FD, Xiao Y, Ohri N, Brockway KD, Piper JW, Nelson AS. What is the best way to contour lung tumors on PET scans? Multiobserver validation of a gradient-based method using a NSCLC digital PET phantom. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):1164-71. doi: 10.1016/j.ijrobp.2010.12.055. Epub 2011 Apr 29. PMID 21531085